CLINICAL TRIAL: NCT00710762
Title: A Randomised Placebo-Controlled Phase II Study of Continuous Maintenance Treatment With BIBF 1120 Following Chemotherapy in Patients With Relapsed Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Model: Parallel | Purpose: Prevention
Other Study IDs: 1199.9; EUDRACT2005-002427-14; NCT00370175 (obsolete NCT alias)
Record Dates: First submitted 2008-07-03; First posted 2008-07-04 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-07

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — nintedanib

ARMS (2):
- BIBF1120 (Experimental)
  Interventions: Drug: BIBF1120
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIBF1120
  Arms: BIBF1120
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to estimate the Progression Free Survival Rates (PFS) of patients with relapsed ovarian cancer after 9 months of continuous treatment with either BIBF 1120 or matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with histologically confirmed advanced ovarian carcinoma, fallopian tube carcinoma or primary peritoneal cancer of serous type with recurrent disease and who responded to 2nd, 3rd or 4th line chemotherapy. Response is defined as either a confirmed decline in CA125 of at least 50% from the pre-treatment value or an Objective Response, i.e. a Partial Response (PR) or Complete Response (CR) according to the RECIST criteria in patients with measurable disease.
* Treatment-free interval of < 12 months since commencing prior treatment regimen for relapsed ovarian cancer.
* Full recovery from all therapy related toxicities of previous chemotherapy and or radiotherapy or recovery in as much as no further improvement may be expected by the investigator.
* Age > 18 years.
* Life expectancy of at least 3 months.
* ECOG Performance Score < 2.
* Adequate hepatic function: total bilirubin 26µmol/L, ALT and/or AST 1.5x upper limit of normal (ULN). INR, Prothrombin time (PT) and partial thromboplastin time (PTT): maximum 50% deviation from normal limits.
* Adequate renal function: serum creatinine 1.5 x ULN.
* Absolute neutrophil count (ANC) >1.5 x 109l, Platelets > 100 x 109/l, Haemoglobin > 9.0 g/dl.
* Written informed consent consistent with ICH-GCP guidelines.
* Minimum time elapsed since last chemotherapy (including hormonal treatment other than Hormone Replacement Therapy [HRT]) or immunotherapy and the first administration of BIBF 1120 must be more than 4 but less than 8 weeks.

Exclusion Criteria:

* Serious illness or concomitant non-oncological disease such as neurologic, psychiatric, infectious disease or active ulcers (gastro-intestinal tract, skin) or laboratory abnormality that may increase the risk associated with study participation or study drug administration and in the judgment of the investigator would make the patient inappropriate for entry into the study.
* Major injuries and/or surgery within past 4 weeks with incomplete wound healing or bone fracture and planned surgical procedures during the study period.
* Hypersensitivity to BIBF 1120 or the excipients of the study drug.
* Significant cardiovascular diseases (i.e. uncontrolled hypertension, unstable angina, history of infarction within past 9 months, congestive heart failure > NYHA II).
* History of haemorrhagic or thrombotic event in the past 12 months. Known inherited predisposition to bleeds or to thrombosis.
* Patients who require full-dose anticoagulation.
* Gastrointestinal disorders or abnormalities that would inhibit absorption of the study drug.
* Brain metastases or leptomeningeal disease.
* Treatment with other investigational drugs or participation in another clinical trial within the past four weeks before start of therapy or concomitantly with this trial.
* Chemo-, radio-, or immunotherapy within the past four weeks prior to treatment with the trial drug.
* Patients unable to comply with the protocol.
* Active alcohol or drug abuse.
* Other documented malignancy with the exception of non-melanomatous skin cancer within the past 5 years.
* Patients who are not clinically sterile.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2006-03; Primary Completion 2008-09 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (11):
- United Kingdom (11):
  - 1199.9.4413 Boehringer Ingelheim Investigational Site, Burton-on-Trent
  - 1199.9.4412 Boehringer Ingelheim Investigational Site, Cambridge
  - 1199.9.4407 Boehringer Ingelheim Investigational Site, Creigiau, Cardiff
  - 1199.9.4410 St James's University Hospital, Leeds
  - 1199.9.4401 Boehringer Ingelheim Investigational Site, London
  - 1199.9.4404 Boehringer Ingelheim Investigational Site, London
  - 1199.9.4409 Boehringer Ingelheim Investigational Site, London
  - 1199.9.4411 Boehringer Ingelheim Investigational Site, London
  - 1199.9.4406 Boehringer Ingelheim Investigational Site, Manchester
  - 1199.9.4402 Boehringer Ingelheim Investigational Site, Northwood
  - 1199.9.4405 Boehringer Ingelheim Investigational Site, Sutton

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 89 patients were enrolled and 84 patients were randomised for this study.
Groups:
- Nintedanib: Patients were treated with 250mg nintedanib twice daily
- Placebo: Patients were treated with matching placebo twice daily
Period: Overall Study
Arm/Group | Nintedanib | Placebo
Started | 44 | 40
Completed | 5 | 0
Not Completed | 39 | 40
Not completed — Progressive disease | 27 | 30
Not completed — Adverse Event other disease worsening | 2 | 1
Not completed — Other Adverse Event | 7 | 7
Not completed — Lost to Follow-up | 1 | 0
Not completed — Reason other than listed above | 2 | 2

BASELINE CHARACTERISTICS:
Population: Treated set consist of all patients who received at least 1 dose of nintedanib or placebo.
  Note: 43 patients were included in the analyses instead of 44 patients in nintedanib arm as one patient was excluded after drug administration due to important protocol violation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nintedanib | Placebo | Total
Number analyzed (Participants) | 43 | 40 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (9.5) | 61.3 (9.1) | 59.8 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 40 | 83
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: PFS Rate at 36 Weeks (After 9 Months)
Description: The rate (probability) of being progression free at Week 36. Progression Free Survival (PFS) was defined according to RECIST version 1.0 from the time of first study drug administration to the first time of either objective tumour progression, the appearance of ≥1 new tumour lesion(s), occurrence or significant progression of malignant ascites, tumour related death, or the time when patients were censored at last known follow up. The rate is the Kaplan-Meier estimated percent probability.
Time Frame: 36 weeks (after 9 months)
Population: Treated set.
Measure: Number (95% Confidence Interval); unit: percent probability of PFS
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 43 | 40
percent probability of PFS | 15.6 [3.8 to 27.3] | 2.9 [0.0 to 8.4]

2. Secondary Outcome: PFS Rate at 12 Weeks (After 3 Months) and 24 Weeks ( After 6 Months)
Description: The rate (probability) of being progression free at Week 12 and Week 24. Progression Free Survival (PFS) was defined according to RECIST version 1.0 from the time of first study drug administration to the first time of either objective tumour progression, the appearance of ≥1 new tumour lesion(s), occurrence or significant progression of malignant ascites, tumour related death, or the time when patients were censored at last known follow up. The rate is the Kaplan-Meier estimated percent probability.
Time Frame: 12 weeks (after 3 months) and 24 weeks ( after 6 months)
Population: Treated set
Measure: Number (95% Confidence Interval); unit: percent probability of PFS
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 43 | 40
percent probability of PFS
  at 24 weeks ( after 6 months) | 26.7 [12.5 to 40.8] | 17.3 [5.2 to 29.4]
  at 12 weeks (after 3 months) | 45.3 [29.5 to 61.2] | 46.2 [30.5 to 61.8]

3. Secondary Outcome: Time to Tumour Progression
Description: Time to Tumour Progression according to RECIST version 1.0 , CA-125 (ovarian tumour marker) levels and RECIST + CA-125 levels.
  For CA-125, progressive disease was defined on the basis of progressive serial elevations of CA-125 according to the following criteria:
  Patients with elevated CA-125 pre-treatment and normalisation of CA-125 had to show evidence of CA-125 levels ≥2 x ULN on 2 occasions at least 1 week apart. or Patients with elevated CA-125 pre-treatment that never normalised had to show evidence of CA-125 levels ≥2 x the nadir value on 2 occasions at least 1 week apart. or Patients with CA-125 in the normal range pre-treatment had to show evidence of CA-125 levels ≥2 x ULN on 2 occasions at least 1 week apart.
  Composite (RECIST+CA-125) endpoint is the RECIST progressive disease (PD) if it occurred or the CA-125 PD if it occurred in the absence of RECIST PD.
Time Frame: 9 months
Population: Treated set
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 43 | 40
days
  according to RECIST and CA-125 | 83.00 [78.0 to 149.0] | 84.00 [78.0 to 87.0]
  according to CA-125 | 85.00 [79.0 to 149.0] | 86.00 [67.0 to 113.0]
  according to RECIST | 143.0 [82.0 to 175.0] | 85.0 [78.0 to 89.0]

4. Secondary Outcome: Time to Death
Description: This end point was not determined as no patients died during the trial.
Time Frame: 9 months
Population: This endpoint could not be calculated as no patients died.
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Incidence and Intensity of Adverse Events With Grading According CTCAE
Description: Incidence and intensity of Adverse Events with grading according to the Common Terminology Criteria for Adverse Events (CTCAE version 3.0).
Time Frame: First drug administration until 28 days after last drug administration,up until 309 days
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 43 | 40
percentage of participants
  CTCAE grade 1 | 2.3 | 25.0
  CTCAE grade 2 | 34.9 | 42.5
  CTCAE grade 3 | 53.5 | 25.0
  CTCAE grade 4 | 7.0 | 2.5
  CTCAE grade 5 | 0.0 | 0.0

6. Secondary Outcome: Clinical Relevant Abnormalities for Laboratory Parameters
Description: Clinical Relevant Abnormalities for laboratory parameters. Any new or clinically relevant worsening of baseline conditions was reported as Adverse Events.
Time Frame: First drug administration until 28 days after last drug administration, up until 309 days
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 43 | 40
Percentage of participants
  Alanine aminotransferase increased | 37.2 | 7.5
  Gamma-glutamyltransferase increased | 30.2 | 2.5
  Aspartate aminotransferase increased | 25.6 | 2.5
  Blood alkaline phosphatase increased | 7.0 | 5.0
  Blood lactate dehydrogenase increased | 4.7 | 0.0
  Blood alkaline phosphatase | 0.0 | 2.5
  Blood alkaline phosphatase abnormal | 2.3 | 2.5
  Lymphocyte count decreased | 0.0 | 2.5
  Vitamin B12 decreased | 0.0 | 2.5
  Alanine aminotransferase abnormal | 2.3 | 0.0
  Blood lactate dehydrogenase abnormal | 2.3 | 0.0
  Gamma-glutamyltransferase abnormal | 2.3 | 0.0
  Neutrophil count decreased | 2.3 | 0.0
  White blood cells urine positive | 2.3 | 0.0
  Blood pressure increased | 0.0 | 2.5
  Electrocardiogram T wave amplitude decreased | 0.0 | 2.5
  Liver function test abnormal | 2.3 | 0.0

ADVERSE EVENTS:
Time Frame: First drug administration until 28 days after last drug administration, up until 309 days
Arm/Group | Nintedanib | Placebo
Serious Adverse Events (participants affected / at risk) | 14/43 | 10/40
Other Adverse Events (participants affected / at risk) | 42/43 | 37/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib (N=43) | Placebo (N=40)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 2
Ascites (Gastrointestinal disorders) | 6 | 5
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 10 | 0
Pyrexia (General disorders) | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Delusion (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib (N=43) | Placebo (N=40)
Tinnitus (Ear and labyrinth disorders) | 3 | 1
Abdominal distension (Gastrointestinal disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 23 | 15
Constipation (Gastrointestinal disorders) | 9 | 11
Diarrhoea (Gastrointestinal disorders) | 33 | 14
Dyspepsia (Gastrointestinal disorders) | 3 | 1
Flatulence (Gastrointestinal disorders) | 5 | 4
Nausea (Gastrointestinal disorders) | 32 | 13
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 1
Stomatitis (Gastrointestinal disorders) | 5 | 1
Vomiting (Gastrointestinal disorders) | 23 | 9
Fatigue (General disorders) | 12 | 11
Oedema peripheral (General disorders) | 1 | 3
Infection (Infections and infestations) | 3 | 1
Nasopharyngitis (Infections and infestations) | 6 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 3
Urinary tract infection (Infections and infestations) | 4 | 4
Alanine aminotransferase increased (Investigations) | 16 | 3
Aspartate aminotransferase increased (Investigations) | 10 | 1
Gamma-glutamyltransferase increased (Investigations) | 12 | 1
Anorexia (Metabolism and nutrition disorders) | 11 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2
Dizziness (Nervous system disorders) | 4 | 4
Headache (Nervous system disorders) | 6 | 4
Lethargy (Nervous system disorders) | 4 | 4
Neuropathy peripheral (Nervous system disorders) | 0 | 3
Paraesthesia (Nervous system disorders) | 1 | 4
Anxiety (Psychiatric disorders) | 2 | 4
Insomnia (Psychiatric disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 6
Rash (Skin and subcutaneous tissue disorders) | 3 | 5
Hot flush (Vascular disorders) | 3 | 3
Hypertension (Vascular disorders) | 5 | 2

LIMITATIONS AND CAVEATS:
Data from all randomised patients collected upto NOV'08 were included in all above sections,unless stated otherwise.5 patients continued on BIBF1120 after database lock(DBL)-NOV'08 upto Mar'14,but due to limited data no further analyses were done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.